CLINICAL TRIAL: NCT03076593
Title: GAPcare: The Geriatric Acute and Post-acute Care Coordination Program - Pilot Survey
Brief Title: GAPcare Fall Prevention Pilot Survey
Status: Completed | Type: Observational
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UEMF0010
Record Dates: First submitted 2017-03-02; First posted 2017-03-10 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Fall
Keywords: geriatric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exposure: Fall — Participants will be asked about prior falls

SUMMARY:
GAPcare (Geriatric Acute & Post-acute Care Coordination Program for Fall Prevention) is an early stage investigation that surveys older adults who present to the Emergency Department for any illness to determine the feasibility of an Emergency Department (ED)-based multidisciplinary intervention for preventing recurrent falls in older adults. In this observational study, older adults will be approached during routine clinical care in the ED and asked about prior falls, prior experiences having falls treated in the inpatient and outpatient setting, and the investigators will solicit feedback on potential improvement to care in the ED setting for falls.

ELIGIBILITY:
Study inclusion criteria for GAPcare

* Adult 65 years-old or older
* Able to communicate in English
* No cognitive impairment (≥4 on SIS)

Exclusion criteria

• Unable to give informed consent due to intoxication or altered mental status

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults presenting to the Emergency Department at Rhode Island Hospital for any indication
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of enrollment | at study enrollment
  The investigators will assess the number of patients who were screened and enrolled at the study site

SECONDARY OUTCOMES:
Type of preventative services offered after a prior fall | at study enrollment
  Participant will be asked what services they were provided after prior falls.
Satisfaction with prior Emergency Department evaluations after a fall using a likert scale | at study enrollment
  Participant will be asked about their satisfaction with prior fall assessments in the ED.
Feedback on prior fall evaluations | at study enrollment
  Participants will give free-text feedback on their perception of the quality of prior outpatient and inpatient fall care

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Goldberg, MD, Principal Investigator — Rhode Island Hospital, Brown University
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No